CLINICAL TRIAL: NCT05276193
Title: GamReg Sweden - Quality Register for Gambling and Gaming Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: GamReg Sweden
Record Dates: First submitted 2022-02-11; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Gambling Disorder; Gaming Disorder
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational health care register - no applicable intervention at present — Observational health care register - no applicable intervention at present

SUMMARY:
This is a quality register for the monitoring of clinical assessment and treatment for gambling disorder and gaming disorder in Swedish health care.

This register is held by Region Skåne, the health care organization of Skåne in southern Sweden, and administered by Register center South, which is associated with health care services in the southern regions of Sweden (the establishment of quality registers in Swedish health care relies upon a national legislation). Quality registers by themselves do not represent formal research projects. However, future research projects can use quality registers, such as the present one, as a data source for future research projects in case they are approved by an ethics authority.

Clinical study variables collected in the register include the following (examples):

* gender, age, occupation, living conditions
* if applicable, types of gambling associated with the treatment needs
* if applicable, type of problematic video gaming
* type of referral to the present treatment contact
* treatment history in psychiatry, social services, enforcement agency
* history of suicidal behavior
* alcohol and drugs problems requiring assessment or treatment
* violence victimization
* type of treatment provided to the patient

ELIGIBILITY:
Inclusion Criteria:

* All patients assessed and treated at units where treatment of problem gambling or problem gaming is provided

Exclusion Criteria:

* Patients who - in a standardized opt-out procedure (following standard of national regulation for quality registers) - refuse participation in the quality register

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All included subjects.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment uptake | 1 year
  Number of patients treated (assessed annually)
Characteristics of treatment-seeking patients | 1 year
  Characteristics of treatment-seeking patients (socio-demographic and mental health co-morbidities), assessed annually
Distribution of treatment methods provided (assessed annually) | 1 year
  Distribution of treatment methods provided (cognitive-behavioral therapy, motivational interviewing, psycho-dynamic treatment, medication, etc, assessed annually)

CONTACTS AND LOCATIONS:
Locations (1):
- Malmö Addiction Center, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hakansson A, Akesson G. GamReg Sweden-Protocol for a systematic cohort data collection for improved clinical knowledge in specialized gambling disorder treatment. Front Psychiatry. 2022 Sep 12;13:894532. doi: 10.3389/fpsyt.2022.894532. eCollection 2022. PMID 36172517
- See also: Official quality register web page at the register authority (Register Center South, Lund, Sweden), in Swedish — http://rcsyd.se/anslutna-register/gamreg-sweden